CLINICAL TRIAL: NCT03985332
Title: Epidemiological Study on the Evolution of the Rate and Causes of Mortality in Geriatric SRH in the HUS
Brief Title: Evolution of the Rate and Causes of Death in Geriatric SSR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7375
Record Dates: First submitted 2019-04-29; First posted 2019-06-13 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-04

CONDITIONS: Death
Keywords: evolution of the rate; causes of death in geriatric SSR
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In view of the ageing population and the increasing fragility of geriatric patients, it seems interesting to carry out a retrospective epidemiological observational study, on the evolution of the mortality rate and the causes of death in services of suite care and geriatric rehabilitation, in order to apprehend at best the supports, in particular palliative

ELIGIBILITY:
Inclusion Criteria:

* Major patients (≥ 18 years)
* All patients who died during their stay in geriatric SSR between 01/01/2013 and 31/12/2017
* Patients who have not expressed their living refusal to reuse their medical data for research purposes

Exclusion Criteria:

- Refusal on the part of patients of their living to reuse their medical data for research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who died during their stay in geriatric SSR between 01/01/2013 and 31/12/2017
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Study of the different causes of death in geriatric SSR unit | The period from January 1st, 2013 to December 31st, 2017 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Thomas VOGEL, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service Gériatrie, Strasbourg, France